CLINICAL TRIAL: NCT03884322
Title: Self Regulated Physical Activity and Bone Growth Enhancement in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asante Health System (Other)
Responsible Party: Principal Investigator, Barbara Kozol, Barbara Kozol,MS, OTL, staff neonatal occupational therapist, Asante Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AsanteHS
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Prematurity; VLBW - Very Low Birth Weight Infant
Keywords: physical activity; prematurity; bone density; length of stay
MeSH Terms: conditions — Premature Birth; Motor Activity

STUDY DESIGN:
Intervention Model Description: Hypothesis: Premature infants placed in elastic fabric "pods" with opportunity to self initiate exercise pushing against fabric would maintain bone density as well as premature infants receiving traditional joint compression exercises by trained therapists
Masking Description: Masking not possible as obvious which child in pod. Infants were instead matched by age and weight to guarantee uniformity of sample
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prepod Group (Experimental): Premature Infants (31 to 32 weeks gestation on entry to program), healthy who wear a prepod or elastic knit fabric pod with snaps essentially 24 hrs a day with brief breaks for bathing, exams, or parent skin to skin time. The intervention lasts 4 weeks
  Interventions: Other: Prepod
- Control Group (Active Comparator): Premature infants (31 to 32 weeks of age on entry to program), healthy who receive a joint compression exercise program approximately 10 minutes a day 5 days a week. The intervention lasts 4 weeks
  Interventions: Procedure: Joint compression exercises

INTERVENTIONS:
Other: Prepod — the prepod is either a 4 way stretch polyester blend fleece with 8 to 10% lycra, or a 95%cotton5% lycra blend knit. It comes in 4 different sizes to assure a pod that has a conforming but not restricting fit so that the infant is free to stretch in any direction at any time but is loosely held in a position of physiological flexion (the fetal position) when not stretching.
  Arms: Prepod Group
Procedure: Joint compression exercises — Each premature infant enrolled as a control subject received approximately 10 minutes of joint compression exercises provided by a NICU trained physical or occupational therapist 5x a week. The exercises consisted of waking the infant slowly, gently if necessary just before feeding with a simple range of motion stretching program then stabilizing an extremity and applying force distally to proximally for 6 repetitions with a brief pause between each compression.
  Arms: Control Group

SUMMARY:
Premature very low birth weight (VLBW) infants were placed in two groups matched for birth age. The control group received traditional joint compression exercises designed to decrease bone density loss.

Exercises lasted approximately 10 minutes each day 5 days a week. The experimental group were placed in a "prepod", an elastic fabric pod shaped garment or sack on entry into the study and remained in the pod essentially 24 hours a day, with brief breaks for bathing, parental skin to skin experiences,etc. An ultrasound of the left tibia was done on entrance into the study at 31 to 32 weeks gestation and again at completion of the study 4 weeks later. Results showed that experimental infants in pods had slightly less bone density loss than their peers receiving traditional therapy. An incidental finding was that the experimental infants in pods had a significantly shorter length of stay.

DETAILED DESCRIPTION:
During fetal development the developing babe pushes against the uterine wall, often kicking and punching the unfortunate mother, especially during the last few months of pregnancy. The striking out against the resistance of the uterine wall causes joint compression in the arms, legs, and spine and that sensory feedback triggers bone growth. Unfortunately in the premature infant they are robbed of that exercise opportunity and are either splayed out in an incubator trying to copy with movement against gravity or swaddled so that movement isn't really an option. As a result bone density loss occurs in essentially all premature infants and osteopenia or significant loss can be an issue.

Between 1995 and 2008 there was a good deal of work done on identifying the importance of exercise and movement for premature infants. Moyer-Mileur was the leading researcher in the USA who demonstrated that simple exercise programs could prevent or decrease bone density loss. Although there is a shortage of trained therapists to provide these exercises safely they became a fairly common practice by 2010. At about that time the neonatologists at the Asante facility asked to incorporate the exercises into the NICU therapy program and after appropriate training the exercises began.

The Asante NICU is highly developmentally oriented. Infants grow 150 million brain cells an hour during the last few months of pregnancy. Any of the multiple stressors of prematurity can create cortisol and affect that brain growth. For that reason therapists became concerned with the joint compression exercises. While they were good for bone and muscle health the exercises were not always welcomed by the infant. Even the most gentle compassionate therapist is not always welcome if the infant just wants to sleep or be left alone. Therapists sought a system that could provide the needed exercise but in a manner more developmentally appropriate. It took two years of experimenting with different types of materials and different strengths of elasticity before the Prepod design finally evolved. Then the obvious hypothesis was - Will the Prepod be as effective in decreasing bone density loss as the traditional therapy exercises?? After multiple issues replacing originally planned DEXA measurements with safer UTS measurements, the first subjects were enrolled in 2013. Unfortunately in 2015 an issue with the ultrasound machine was identified; the anti-theft anklets the infants wore emitted signals that had corrupted the data. The study needed to be restarted in 2015, removing the anklets prior to measurement. It then proceeded without incident, with expected completion late 2018. At the IRB (Institutional Review Board) review winter of 2017 the overseeing group concluded that the data for length of stay was so compelling that continuing the study wasn't likely to change anything and basically amounted to withholding care from the traditional exercise infants. They ordered early closure of the study, despite the small number of study participants.

ELIGIBILITY:
Inclusion Criteria: 31 to 32 week gestation premature infants AGA (appropriate for gestational age weight) parental consent

Exclusion Criteria: Respiratory disease Low Apgars ( 5 minute less than 4) Syndromes affecting growth SGA (small for gestational age) medication requirements beyond vitamins, iron and caffeine

-

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in bone density | 27 to 28 days
  Infants were divided into two groups - experimental (Prepod) and control (joint compression exercises).
  The infants were measured at 31 to 32 weeks gestation using ultrasound to measure the SOS (speed of sound) through the left tibia at mid point between knee and ankle. They were then remeasured at end of study and the two measurements compared.
Change in length of Stay | 27 to 28 days
  Infants in study were followed to discharge and length of stay from birth to discharge of the two matched groups were compared.

SECONDARY OUTCOMES:
Change of length of stay of all Prepod candidates | 27 to 28 days
  As mentioned in previous documentation the Prepod study began in 2013 but bone density data from 2013 to 2015 had to be discarded due to issues with UTS data corruption. However the infant experience in the Prepod and exercises were identical to those in the final study so length of stay of the combined population was examined.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kozol, MS,OTL, Principal Investigator — Barbara Kozol
Locations (1):
- Rogue Regional Medical Center, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Infant's names were coded on entry into all data tracking for privacy, HIPAA purposes. Individual data and results were not important (beyond assuring they maintained health) as the researcher was looking at overall trends

REFERENCES:
- [Background] Chan GM, Armstrong C, Moyer-Mileur L, Hoff C. Growth and bone mineralization in children born prematurely. J Perinatol. 2008 Sep;28(9):619-23. doi: 10.1038/jp.2008.59. Epub 2008 Jun 12. PMID 18548083
- [Background] Hovi P, Andersson S, Jarvenpaa AL, Eriksson JG, Strang-Karlsson S, Kajantie E, Makitie O. Decreased bone mineral density in adults born with very low birth weight: a cohort study. PLoS Med. 2009 Aug;6(8):e1000135. doi: 10.1371/journal.pmed.1000135. Epub 2009 Aug 25. PMID 19707270
- [Background] Moyer-Mileur L, Luetkemeier M, Boomer L, Chan GM. Effect of physical activity on bone mineralization in premature infants. J Pediatr. 1995 Oct;127(4):620-5. doi: 10.1016/s0022-3476(95)70127-3. PMID 7562289
- [Background] Moyer-Mileur LJ, Brunstetter V, McNaught TP, Gill G, Chan GM. Daily physical activity program increases bone mineralization and growth in preterm very low birth weight infants. Pediatrics. 2000 Nov;106(5):1088-92. doi: 10.1542/peds.106.5.1088. PMID 11061779
- [Background] Vignochi CM, Miura E, Canani LH. Effects of motor physical therapy on bone mineralization in premature infants: a randomized controlled study. J Perinatol. 2008 Sep;28(9):624-31. doi: 10.1038/jp.2008.60. Epub 2008 Jul 17. PMID 18633420
- [Background] Litmanovitz I, Dolfin T, Friedland O, Arnon S, Regev R, Shainkin-Kestenbaum R, Lis M, Eliakim A. Early physical activity intervention prevents decrease of bone strength in very low birth weight infants. Pediatrics. 2003 Jul;112(1 Pt 1):15-9. doi: 10.1542/peds.112.1.15. PMID 12837861
- [Background] Litmanovitz I, Erez H, Eliakim A, Bauer-Rusek S, Arnon S, Regev RH, Sirota G, Nemet D. The Effect of Assisted Exercise Frequency on Bone Strength in Very Low Birth Weight Preterm Infants: A Randomized Control Trial. Calcif Tissue Int. 2016 Sep;99(3):237-42. doi: 10.1007/s00223-016-0145-3. Epub 2016 May 3. PMID 27142078
- [Background] Pereda L, Ashmeade T, Zaritt J, Carver JD. The use of quantitative ultrasound in assessing bone status in newborn preterm infants. J Perinatol. 2003 Dec;23(8):655-9. doi: 10.1038/sj.jp.7211006. PMID 14647163
- [Background] Basu M, Malhotra AS, Pal K, Chatterjee T, Ghosh D, Haldar K, Verma SK, Kumar S, Sharma YK, Sawhney RC. Determination of bone mass using multisite quantitative ultrasound and biochemical markers of bone turnover during residency at extreme altitude: a longitudinal study. High Alt Med Biol. 2013 Jun;14(2):150-4. doi: 10.1089/ham.2012.1042. PMID 23795735